CLINICAL TRIAL: NCT02597010
Title: Dietary Nitrate for Resistant Hypertension: A Randomized, Placebo-controlled, Crossover Trial
Brief Title: A 2 Week, Crossover Trial of Dietary Nitrate in HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University College Dublin (Other); Connolly Hospital Blanchardstown (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Chronic NO3- in HTN
Record Dates: First submitted 2015-01-07; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate rich beetroot juice (Experimental): Concentrated, beetroot juice is a rich source of dietary nitrate.
  Interventions: Dietary Supplement: Dietary nitrate
- Nitrate depleted placebo beetroot juice (Placebo Comparator): Placebo beetroot juice is identical to active beetroot juice in every way except nitrate content.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary nitrate — 140ml of nitrate rich beetroot juice provides 12.9mmol nitrate and will be consumed on a daily basis during the intervention by the study subjects.
  Other Names: Beetroot juice
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Placebo — 140ml of nitrate depleted beetroot juice provides 0.5mmol nitrate and will be consumed on a daily basis during the intervention by the study subjects.
  Other Names: Nitrate depleted beetroot juice
  Arms: Nitrate depleted placebo beetroot juice

SUMMARY:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to decrease systemic blood pressure in multiple populations including newly diagnosed, untreated hypertensives. The additional effect in hypertensives on blood pressure lowering medications is uncertain.

DETAILED DESCRIPTION:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to decrease systemic blood pressure in multiple populations including newly diagnosed, untreated hypertensives. The additional effect in hypertensives on blood pressure lowering medications is uncertain.

The investigators hypothesize that chronic nitrate consumption might decrease blood pressure in hypertensives who are suboptimally controlled on at least one blood pressure medication compared to a placebo beetroot juice.

This study is a randomized, double-blind placebo-controlled, crossover trial. At baseline, mid-point and endpoint ambulatory blood pressure will be assessed in conjunction with demographics and blood draw. After baseline measures, each subject will be randomized to consume nitrate rich beetroot juice for 7 consecutive days when assessments will be repeated followed by 7 days of placebo and endpoint assessments or the converse.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable,
* Uncontrolled hypertension

Exclusion Criteria:

* Pulmonary hypertension
* Active CVD
* Taking vasodilators
* Diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in day ambulatory blood pressure | Day 1, day 15, day 29

SECONDARY OUTCOMES:
Change in plasma nitrate | Day 1, day 15, day 29
Change in 24h ambulatory blood pressure | Day 1, day 15, day 29
Change in night ambulatory blood pressure | Day 1, day 15, day 29
Change in cardiac biomarkers | Day 1, day 15, day 29
  Assessed by serum lipids.
Change in plasma nitrite | Day 1, day 15, day 29
Change in inflammatory biomarkers. | Day 1, day 15, day 29
  Assessed by serum C-reactive protein.